CLINICAL TRIAL: NCT02623673
Title: Simultaneous Therapy With Intravitreal Dexamethasone Implant and Bevacizumab for the Treatment of Macular Edema
Status: Completed | Type: Observational
Sponsor: Retina Clinic, Sao Paulo, Brazil (Other)
Responsible Party: Principal Investigator, Gabriel Costa de Andrade, Gabriel Costa de Andrade, Retina Clinic, Sao Paulo, Brazil
Other Study IDs: Retina CLINIC
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- bevacizumab plus dexamethasone 0.7mg: simultaneous treatment with intravitreal injection of bevacizumab 1.25mg and intravitreal implant of dexamethasone 0.7mg
  Interventions: Drug: simultaneous treatment with intravitreal injection of bevacizumab 1.25mg and intravitreal implant of dexamethasone 0.7mg.

INTERVENTIONS:
Drug: simultaneous treatment with intravitreal injection of bevacizumab 1.25mg and intravitreal implant of dexamethasone 0.7mg.

SUMMARY:
Retrospective cases series is a non-randomized, open-label, single-center investigation (Retina Clinic, São Paulo, Brazil) of patients diagnosed with macular edema secondary to diabetic retinopathy (DME) and retinal vein occlusions who underwent to simultaneous treatment with intravitreal injection of bevacizumab 1.25mg and implant of dexamethasone 0.7mg.

DETAILED DESCRIPTION:
This retrospective cases series is a non-randomized, open-label, single-center investigation (Retina Clinic, São Paulo, Brazil) approved by the Institutional Review Board of Hospital Oftalmológico de Sorocaba/SP, and adhered to the tenets of the Declaration of Helsinki. Were included patients older than 18 years, treated between April 2014 and July 2015, diagnosed with macular edema secondary to diabetic retinopathy (DME) and retinal vein occlusions who underwent to simultaneous treatment with intravitreal injection of bevacizumab 1.25mg (Avastin; Genentech, South San Francisco, CA) and intravitreal implant of dexamethasone 0.7mg (Ozurdex; Allergan, Inc, Irvine, CA).

ELIGIBILITY:
Inclusion Criteria:

* central macular thickness > 300 µm on optical coherence tomography (OCT)
* macular edema secondary to diabetic retinopathy (DME) and retinal vein occlusions

Exclusion Criteria:

* intravitreal anti-VEGF within 6 weeks
* treatment with laser or intravitreal corticosteroids within 3 months of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with macular edema
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Improvement in BCVA | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Clinic / UNIFESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes